CLINICAL TRIAL: NCT04384549
Title: Randomized Controlled Trial Evaluating the Efficacy of Vaccination With Bacillus Calmette and Guérin (BCG) in the Prevention of COVID-19 Via the Strengthening of Innate Immunity in Health Care Workers
Brief Title: Efficacy of BCG Vaccination in the Prevention of COVID19 Via the Strengthening of Innate Immunity in Health Care Workers
Acronym: COVID-BCG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP200462; 2020-001678-31 (EudraCT Number)
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Infection; Viral, Agent as Cause of Disease Classified Elsewhere
Keywords: Vaccinology; Infectiology; COVID-19; Health Workers
MeSH Terms: conditions — Infections; COVID-19 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG Arm (Experimental): One intradermal injection of 0.1 ml of BCG vaccine (AJ Vaccine).Each 0.1 ml vaccine contains between 2 to 8 x 105 colony forming units.
  Interventions: Biological: BCG GROUP
- PLACEBO Arm (Placebo Comparator): One intradermal placebo injection.
  Interventions: Other: PLACEBO GROUP

INTERVENTIONS:
Biological: BCG GROUP — One intradermal injection of 0.1 ml of BCG vaccine (AJ Vaccine).Each 0.1 ml vaccine contains between 2 to 8 x 105 colony forming units.
  Other Names: Experimental GROUP
  Arms: BCG Arm
Other: PLACEBO GROUP — One intradermal injection of 0.1ml NaCl
  Other Names: Control GROUP
  Arms: PLACEBO Arm

SUMMARY:
Healthcare Workers (HCW) are at high risk for COVID-19. In addition to the risk of serious forms among HCW, significant absenteeism due to illness would have dramatic consequences in our ability to fight COVID-19. No coronavirus vaccine is available today and drug treatments are only at the start of clinical evaluation. Available since 1921, the bacillus Calmette and Guérin (BCG) is the most widely used vaccine in the world (> 3 billion doses administered) with an extremely low rate of adverse effects. BCG is indicated for the prevention of tuberculosis (TB), but more recent studies have shown that it also has nonspecific immune properties which may be interesting in the current COVID-19 epidemic. Data in mice and in humans have demonstrated protection conferred by BCG against viral respiratory infections such as influenza. In countries with high endemic TB, BCG decreases the incidence of acute respiratory infections by up to 80%, neonatal BCG vaccination has been shown to greatly reduce the risk of sepsis and of hospitalization of children for reasons other than TB. A recent study conducted in South Africa showed that re-vaccination with BCG in adults reduced the incidence of respiratory infections by 70% compared to unvaccinated controls. Beyond respiratory infections, BCG has also shown protective effects against inflammatory diseases. These non-specific beneficial effects are likely linked to the induction of "trained innate immunity", implying epigenetic and metabolic re-programming of innate immune cells. It is therefore possible that revaccination with BCG could significantly reduce the incidence and severity of COVID-19. Very recent ecological observations indeed suggest an inverse correlation between BCG vaccination coverage and the morbidity and mortality of COVID-19. In this context several trials began in Europe and Australia to evaluate the efficacy of BCG vaccination in populations at risk of exposure (HCW) or severe disease (elderly). This study is aligned with studies carried out in Australia, The Netherlands and Spain. In contrast to these latter studies, virtually all French study participants have been vaccinated in their childhood, since BCG vaccination was mandatory in France in neonates until 2007, and in HCW until recently. Therefore, the French study will be in a unique situation to evaluate the effect of re-vaccination with BCG in the context of BCG priming decades before revaccination.

DETAILED DESCRIPTION:
Randomized, multicenter phase III controlled trial, in 2 parallel arms:

* One group vaccinated with BCG
* One group receiving placebo (0.9 % saline) Randomization in a 1: 1 ratio will be stratified on the center. The study will be proposed to all heath care workers eligible. At screening, the investigator will propose the study to the participant and explain the details by providing an information letter. After signature of the consent, evaluations specific for the study will be undertaken, such as clinical examination, blood sampling, nasopharyngeal sampling in case of clinical signs.

At the inclusion visit, participants corresponding to the inclusion criteria will be randomized to receive BCG or placebo.

Participants will receive a single dose of BCG vaccine (or placebo). The adult dose of BCG vaccine (or placebo) is 0.1 mL injected intradermally over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the upper arm).

Follow-up visits will be done respectively at M3 and M6 and phone contacts between these two visits.

Blood samples will be collected prior to randomization (V0) and at 3 and 6 months to determine exposure to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Where required, swab/blood samples will be taken at illness episodes to assess SARS-CoV-2 infection.

Participants will be followed for 6 months with regular mobile phone text messages 2 times weekly to collect local and general reactions until 30 days after vaccination and during the study to identify and detail COVID-19 infection.

Immunological studies will be conducted at a central Laboratory. Analysis will take place after M6 visits.

A nested study will be carried out on blood samples of 72 study subjects in order to evaluate the impact of COVID-19 on innate immunity. These blood samples will be collected at M6 among 6 groups, each containing 12 study subjects:

* One group of subjects vaccinated with BCG that have remained sero-negative for SARS CoV2
* One group of subjects having received placebo that have remained sero-negative for SARS CoV2
* One group of symptomatic subjects vaccinated with BCG
* One group of symptomatic subjects having received placebo.
* One group without symptoms but sero-positive for SARS CoV2 vaccinated with BCG
* One group without symptoms but sero-positive for SARS CoV2 vaccinated with placebo

ELIGIBILITY:
Inclusion Criteria:

* Individual (Male and female) aged 18 or over.
* Healthcare Worker (medical or non-medical) from hospitals in direct contact with COVID-19 patients.
* Participants must give their written consent before any trial procedure.
* Participants covered by social security regimen (excepting AME).
* Healthy according to the opinion of the investigator.

Exclusion Criteria:

* Has any BCG vaccine contraindication, known allergy to the BCG vaccine or SAE to prior BCG vaccination.
* History of tuberculosis
* People with acquired or innate immunodeficiency.
* People have already been infected with SARS Cov-2 (virological documentation or TDM or seropositive if serology available).
* People who could not commit to follow-up for 6 months.
* People not in good general condition, as assessed by the investigator.
* People included in other clinical trials assessing treatment.
* Pregnant or breastfeeding or positive urine pregnancy at enrolment visit.
* BCG vaccine given within the last year.
* Another live vaccine administered in the month prior to randomization.
* History of anaphylaxis following vaccination.
* Receiving medical treatment that affects the immune response or other immunosuppressive therapy in the last year. These therapies include systemic corticosteroids (more than or equal to 10 mg for more than or equal to 2 weeks), immunosuppressant, biological agents (such as monoclonal antibodies against tumour necrosis factor (TNF)-alpha).
* Another vaccine administered in the month prior to inclusion and randomization.
* Fever > 38°C within the past 24 hours
* People with malignancies (e.g. lymphoma, leukemia, Hodgkin's disease or other tumors of the reticuloendothelial system) or infected with HIV
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Acute severe febrile illness
* Generalized infected skin conditions
* People under legal protection measure (tutorship, curatorship or safeguard measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-02-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of documented COVID-19 among health care workers exposed to SARS CoV2 and vaccinated with BCG compared to placebo. | during the study period of 6 months
  Documented COVID-19, i.e. symptomatic COVID-19 confirmed by either
  * positive nasopharyngeal tests for SARS CoV2
  * and/or by thoracic tomodensitometry compatible with the diagnosis.
  * and/or SARS CoV2 seroconversion

SECONDARY OUTCOMES:
Numbers of COVID-19 patients requiring hospitalization in ICU and O2, artificial ventilation or extracorporal membrane oxygenation, or deaths in BCG-vaccinated health care workers compared to placebo | during the study period of 6 months.
  Participants having developed a severe form of COVID-19, as defined by the necessity for hospitalization in ICU and O2 or artificial ventilation, or extracorporeal membrane oxygenation, or death
Incidence of asymptomatic SARS CoV2 seropositive subjects among BCG-vaccinated health care workers compared to placebo. | during the study period of 6 months.
  Participants with seroconversion during the study, without symptoms related to COVID-19
Incidence of subjects with any respiratory infection among BCG-vaccinated health care workers compared to placebo. | during the study period of 6 months.
  Participants presenting any kind of respiratory infection due to any cause
Numbers of sick days and numbers of sick leaves among BCG-vaccinated health care workers compared to placebo. | during the study period of 6 months
  Numbers of sick days and number of sick leaves
Numbers of subjects with BCG-related advers events among BCG-vaccinated health care workers compared to placebo. | 30 days after BCG revaccination
  Local and general events following BCG revaccination after BCG revaccination
Numbers and intensity of changes in innate immune markers after SARS CoV2 infection among BCG-vaccinated health care workers compared to placebo. | during the study period of 6 months.
  Potentially modified markers of innate immunity upon SARS CoV-2 infection to be identified

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, Professor, Principal Investigator — Assitance Publique-Hôpitaux de Paris; Camille LOCHT, Professor, Study Director — Institut Pasteur de Lille
Locations (1):
- I-REIVAC/CIC 1417 Cochin Hospital, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moorlag SJCFM, Arts RJW, van Crevel R, Netea MG. Non-specific effects of BCG vaccine on viral infections. Clin Microbiol Infect. 2019 Dec;25(12):1473-1478. doi: 10.1016/j.cmi.2019.04.020. Epub 2019 May 2. PMID 31055165
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] Kowalewicz-Kulbat M, Locht C. BCG and protection against inflammatory and auto-immune diseases. Expert Rev Vaccines. 2017 Jul;16(7):1-10. doi: 10.1080/14760584.2017.1333906. Epub 2017 May 30. PMID 28532186
- [Background] Netea MG, Dominguez-Andres J, Barreiro LB, Chavakis T, Divangahi M, Fuchs E, Joosten LAB, van der Meer JWM, Mhlanga MM, Mulder WJM, Riksen NP, Schlitzer A, Schultze JL, Stabell Benn C, Sun JC, Xavier RJ, Latz E. Defining trained immunity and its role in health and disease. Nat Rev Immunol. 2020 Jun;20(6):375-388. doi: 10.1038/s41577-020-0285-6. Epub 2020 Mar 4. PMID 32132681
- See also: Miller A, et al. 2020. Correlation between universal BCG vaccination policy and reduced morbidity and mortality for COVID-19: an epidemiological study. — https://doi.org/10.1101/2020.03.24.20042937